CLINICAL TRIAL: NCT04821648
Title: A Study of the Safety, Tolerability, and Clinical Pharmacology of Subcutaneous Rjv001 in Adult Subjects Undergoing Abdominoplasty
Brief Title: RJV001 Study in Adults Receiving Abdominoplasty
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rejuven Dermaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Joseph Gimbel, MD, Chief Medical Officer, Rejuven Dermaceutical Co., Ltd.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RJV001-PH1-01
Record Dates: First submitted 2021-03-25; First posted 2021-03-29 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Submental Fat (SMF); Double Chin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dosage group A (Experimental): Dosage group A will consist of 6 subjects, 1:1:1 (A1:A2:A3 below):
  A1: 0.04 mg/injection; A2: 0.075 mg/injection; A3: 0.15 mg/injection Two subjects will be dosed in the area scheduled for resection with 5 injections of the lowest of the 3 RJV001 test article strengths (i.e., 0.04 mg/injection); the two subjects will also be dosed with a single injection of vehicle in the area scheduled for resection for a total of 6 injections. At the conclusion of a given test article dose group, if tolerated, enrollment will continue to the next higher dose after approval to advance based upon an interim safety review. This same process will be repeated for the 0.075 mg/injection dose with 2 additional subjects. Assuming the interim safety review for the mid dose (i.e., 0.075 mg/injection) is deemed acceptable, the 2 final subjects will be treated with the high dose (0.15 mg/injection).
  Interventions: Drug: RJV001; Drug: Placebo
- Dosage group B (Experimental): Dosage group B will consist of 3 subjects (if only 1 dose from Dosage group A is well tolerated) or 6 subjects (if 2 doses from Dosage group A are well tolerated), randomized 1:1 (B1:B2 below).
  B1: RJV001 Solution for Injection, Dose 1 B2: RJV001 Solution for Injection, Dose 2 Subjects will be dosed with 1 RJV001 test article (i.e., one of the 2 highest concentrations of RJV001 doses that were well tolerated in Dosage group A, referred to as Dose 1 and Dose 2). Up to 13 injections (12 active and 1 vehicle) will be administered in an open label manner in the area scheduled for resection. If tolerated, enrollment will continue to Dosage group C after approval to advance based upon an interim safety review.
  Interventions: Drug: RJV001; Drug: Placebo
- Dosage group C (Experimental): Dosage group C will consist of 3 subjects (if only 1 dose from dosage group B is well tolerated) or 6 subjects (if 2 doses from Dosage group B are well tolerated), randomized 1:1 (C1:C2 below).
  * C1: RJV001 Solution for Injection, Dose 1
  * C2: RJV001 Solution for Injection, Dose 2 Subjects will be dosed with 1 RJV001 test article (i.e., one of the 2 highest concentrations of RJV001 doses that were well tolerated in Cohort B, referred to as Dose 1 and Dose 2). Up to 31 injections (30 active and 1 vehicle) will be administered in an open-label manner in the area scheduled for resection.
  Interventions: Drug: RJV001; Drug: Placebo

INTERVENTIONS:
Drug: RJV001 — Subcutaneous injection in the abdomen
Drug: Placebo — The placebo formulation has the same shape, color, and qualitative composition as the RJV001 freeze dried powder, with the exception that RJV001 drug substance has been removed. For each cohort group, a placebo will be injected in a single site in the same area as the treatment.

SUMMARY:
In this study, we are testing a new drug against submental fat (SMF), which is characterized with the accumulation of fat under the chin that often appears as a "double chin". The 2018 American Society for Dermatologic Surgery Consumer Survey on Cosmetic Dermatologic Procedures indicated that 73% of respondents were bothered by "excess fat under the chin/neck". This condition of loose or sagging skin under the chin may affect facial symmetry and attractiveness, which can lead to social embarrassment and a negative self-image in many patients.

There is an insufficiency in effective drugs against SMF and double chin. Although an injectable small molecule can be used for improvement of double chin, but its side effects are evident and its cost is high. As such, there remains a real need to develop a cost-effective method to improve appearance of SMF and double chin.

DETAILED DESCRIPTION:
The therapies directed against adipocytes represent a novel therapeutical approach for improving the appearance of double chin. Furthermore, these treatments would optimally work by novel mechanisms so that the enhanced adverse effects at injection sites will not limit their use. Our studies suggest that RJV001 may fulfill these requirements.

Adipocytes are attached to an extracellular matrix (ECM) that mainly consists of a collagen network, the degradation of which may induce apoptosis of adipocytes, leading to the improvement of the double chin's appearance. Collagenases are enzymes that break the peptide bonds in collagen; collagenase-induced destruction of the collagen network may lead to improvement in the appearance of the double chin.

Rejuven is currently developing RJV001 for improving the appearance of moderate to severe convexity or fullness-associated SMF in adults. RJV001 is a mutant recombinant collagenase of Clostridium histolyticum, which contains one amino acid difference. This amino acid is in the active center and preclinical studies showed that Kcat of RJV001 was significantly lower than that of the wild type enzyme, but Km of RJV001 was close to that of the wild type. Preclinical studies conducted by Rejuven also demonstrated that RJV001 can still effectively induce lipolysis of fat tissue and that the decreased bioactivity may have the benefit of decreased adverse effects.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a male or non-pregnant female 18-65 years of age.
2. Subject has provided written informed consent.
3. Females must be post-menopausal , surgically sterile , or use an effective method of birth control. , Women of childbearing potential (WOCBP) must have a negative urine pregnancy test (UPT) at Visit 1/Screening and Visit 2/Baseline.
4. Subject is scheduled on a specific date to undergo abdominoplasty and meets all pre-operative requirements, in the opinion of the investigator.
5. Subject is willing to undergo test article injections as directed, comply with study instructions, and commit to all follow-up visits for the duration of the study.
6. Subject, in the investigator's opinion, is in good general health and free of any disease state or physical condition that might impair evaluation of the test article injection sites or expose the subject to an unacceptable risk by study participation.

Exclusion Criteria:

1. Subject is pregnant, lactating, or is planning to become pregnant during the study.
2. Subject has a significant active systemic or localized abdominal infection.
3. Subject has any medical condition that affects clotting and/or platelet function (e.g., thromboembolic disease, clotting factor deficiencies such as hemophilia).
4. Subject is taking any medications that affect clotting and/or platelet function. This includes, but is not limited to, nonsteroidal anti-inflammatory medications (including low dose aspirin for prophylaxis), heparin (including low molecular weight heparin), Coumadin, and factor Xa agents such as Clopidogrel bisulfate (Plavix) and apixaban (Eliquis), etc. The use of such medications is precluded within 7 days prior to Visit 2/Baseline.
5. Subject is immunocompromised, in the opinion of the investigator, based on their medical condition (e.g., positive for human immunodeficiency virus, malignancy), medication use, or other factors.
6. Subject has any clinically significant medical abnormality or chronic disease of the cardiovascular, gastrointestinal, respiratory (e.g., chronic obstructive pulmonary disease), hepatic, or renal systems. This includes conditions (e.g., gastrointestinal surgery) that may interfere with metabolism or excretion.
7. Subject is currently enrolled in an investigational drug or device study.
8. Subject has used an investigational drug or investigational device treatment within 30 days prior to Visit 2/Baseline.
9. Subject has a history of sensitivity to RJV001, other collagenases, or any of the other ingredients in the test articles.
10. Subject is known to be noncompliant or is unlikely to comply with the requirements of the study protocol (e.g., due to alcoholism, drug dependency, mental incapacity) in the opinion of the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2021-12-16 (Actual)

PRIMARY OUTCOMES:
Local and systemic adverse events following administration of RJV001 | 30 minutes
  * Necrosis
  * Thrombosis
  * Ischemia
  * Gangrene
  * Injection site discoloration
  * Allergic dermatitis
  * Neovascularization
  * Nerve injury
  * Pain

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Gimbel, M.D., Principal Investigator — Arizona Research Center
Locations (1):
- Study site: Arizona Research Center, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Asds consumer survey on cosmetic dermatologic procedures: American Society for Dermatological Surgery; 2018. (Available from: https://www.asds.net/Portals/0/PDF/consumer-survey-2018-infographic.pdf.)
- [Result] Schlessinger J, Weiss SR, Jewell M, Narurkar V, Weinkle S, Gold MH, Bazerkanian E. Perceptions and practices in submental fat treatment: a survey of physicians and patients. Skinmed. 2013 Jan-Feb;11(1):27-31. PMID 23540074
- [Result] Mukherjee A. Pharmacology review(s) of xiaflex. 2009.